CLINICAL TRIAL: NCT07234617
Title: Evaluating Public Policy: A Case Study of the Green Prescription POLVERT (Green Policy - Evaluation and Results)
Brief Title: Public Policy Evaluation: the Case of the Green Prescription
Acronym: POLVERT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 9588
Record Dates: First submitted 2025-11-14; First posted 2025-11-18 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Pregnancy
Keywords: Pesticides; organic vegetables

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (No Intervention): Vegetable consumption according to habits
- Intervention (Experimental): Consumption of organic vegetables
  Interventions: Behavioral: Consumption of organic vegetables

INTERVENTIONS:
Behavioral: Consumption of organic vegetables — Consumption of organic vegetables or non-organic for control group (according to their usual habits) for 2 weeks
  Arms: Intervention

SUMMARY:
Numerous studies have highlighted the harmful effects of pesticide exposure during the prenatal period. Food is one of the main vectors of exposure to pesticides, particularly glyphosate, which is the most widely used herbicide. Observational studies have highlighted their effects on health, but few interventional studies have been conducted to identify effective interventions to reduce or eliminate environmental risks. In 2022, the City of Strasbourg implemented the "Ordonnance Verte" (Green Prescription) program, giving all pregnant women in the city access to a weekly basket of organic and local vegetables for several months, as well as awareness-raising workshops on endocrine disruptors and healthy eating. The objective of this study is to assess whether this type of program reduces pregnant women's exposure to pesticides compared to women who continue to eat according to their usual habits. If conclusive, this type of assessment would play a key role in facilitating the rollout of similar initiatives on a larger scale and protecting the health of pregnant women and future children.

ELIGIBILITY:
Inclusion Criteria:

* Be a woman
* Be less than 32 weeks pregnant
* Be registered with the "Ordonnance Verte" program
* Have agreed, when registering for the program, to be contacted by a research team
* Be affiliated with a social security system or be a beneficiary of such a system.
* Be fluent in French.
* Be over 18 years of age
* Be able to understand the objectives and risks associated with the research and give dated and signed informed consent
* Have a telephone and internet access

Exclusion Criteria:

* Participation in a study on nutrition or any other studies likely to affect exposure to the compounds under investigation
* Inability to provide informed consent (difficulties in understanding on the part of the pregnant woman, etc.)
* Being under judicial protection
* Being under guardianship or conservatorship
* Working in the agricultural sector (farmer, employee, apprentice)
* Living with someone who works in the agricultural sector (farmer, employee, apprentice)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 210 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Change in urinary pesticide concentrations over the two-week study period in the intervention group | Day 0 and at 2 weeks
  Measured as the difference in pesticide levels before and after the intervention
Difference in urinary pesticide concentrations between the two groups | Day 0 and at 2 weeks
  Measured as the difference in pesticide levels in intervention vs. control groups

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France

IPD SHARING:
Plan to Share IPD: No